CLINICAL TRIAL: NCT04840316
Title: INcidence of PostOperative Delirium Incidence in Surgical Patients: an Observational Cohort Study in New Zealand
Acronym: INPOD-NZ
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Auckland City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: A+ 9133
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-05

CONDITIONS: Delirium Confusional State; Complication,Postoperative
Keywords: Anesthesia; Delirium; Incidence; Cognitive decline
MeSH Terms: conditions — Confusion; Postoperative Complications; Delirium; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post operative: Nil Intervention - observational cohort study

SUMMARY:
As the population of older adults increases, so too with the number of older adult patients that present for anesthesia and surgery. The development of delirium following surgery has some significant potential effects on patient outcomes; however, POD is often under diagnosed. Some studies reported that more than 50% of patients with delirium were undiagnosed by clinical teams. POD is associated with cognitive decline, increased hospital length of stay, discharge to institutional care, mortality and higher healthcare costs. POD contributes significantly to healthcare inefficiency; a diagnosis of POD is estimated by the Australian Commission on Quality and Safety in Healthcare to cost an additional $27,791 AUD. The incidence of POD reported in clinical trials depends on the risk profile of the study population, the frequency and duration of delirium assessments as well as the surgical procedure. Reported incidence may also vary due to the presence of high-risk pathways involving multi-specialty management and intervention. POD may present as either hyperactive or hypoactive subtypes, the latter being more difficult to detect.

There are few reports on the incidence of POD in New Zealand national level datasets, with single centre studies primarily looking at in-hospital delirium and demonstrating an incidence of 11.2 to 29% on mixed and/or medical wards. A review of elderly patients with neck-of-femur fractures found the incidences of POD to be as high as 39%. The current data suggests a significant level of morbidity due to POD in New Zealand hospitals, however there is lack of national level data in the surgical population; which is crucial for establishing demographic and regional need for effective intervention.

ELIGIBILITY:
Eligible patients include those aged 18 years or over undergoing a surgical procedure in any of 71 public or private hospitals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participant patients will have been assigned procedure codes for surgery and anaesthesia. Patients who had multiple procedures during an episode of care will have each procedure and relevant postoperative course analysed. Patients were excluded if the procedure was performed under local anaesthesia infiltration. Procedures performed under regional or neuraxial techniques will be included in the analysis.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2021-06-30 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | January 1st 2007 to December 31st 2016
  Clinical outcomes are coded by trained clinical coders at each individual hospital and reported to the Ministry of Health as per standard practice. Delirium will be defined by the ICD-9 and ICD-10 coding of delirium as an outcome [12]. POD will be defined as the presence of an ICD-9 or ICD-10 delirium code following surgery until seven days postoperatively or discharge, whichever occurs earlier. If a patient received multiple eligible operations during the captured time frame, each surgical event postoperatively will be analysed individually.

CONTACTS AND LOCATIONS:
Locations (1):
- Auckland City Hopsital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No
As an observational study of encrypted data from the national data set there is no plan to provide individual participant data.